CLINICAL TRIAL: NCT05350358
Title: A Retrospective Patient Registry on the Long-Term Performance of the Dialine II® Vascular Graft Prosthesis Used in Open Vascular Surgery
Brief Title: LeMaitre® CARDIAL Dialine II Post Market Study
Acronym: Dialine II®
Status: Completed | Type: Observational
Sponsor: Geprovas (Network)
Collaborators: LeMaitre Vascular (Industry)
Responsible Party: Sponsor
Other Study IDs: DLN-41-001
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Vascular Aneurysm; Vascular Occlusive Disease; Artery Injury
Keywords: Vascular prosthesis; Aneurysm; Occlusion; Arterial reconstruction
MeSH Terms: conditions — Aneurysm; Bites and Stings

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have undergone surgical treatment with LeMaitre Cardial Dialine II: Subject who has undergone surgical treatment for the replacement or bypass in aneurysmal and/or occlusive diseases and for arterial reconstruction in patients requiring systemic heparinization with LeMaitre Cardial Dialine II.
  Interventions: Device: LeMaitre Cardial Dialine II

INTERVENTIONS:
Device: LeMaitre Cardial Dialine II — Surgical treatment for the replacement or bypass with LeMaitre Cardial Dialine II

SUMMARY:
This clinical study will capture clinical data specific to the performance and safety of the LeMaitre® CARDIAL Dialine II. It is a retrospective, monocenter, post-market safety and performance study. Following the new MDR regulation, this study will allow the clinical data of the prosthesis to be completed in order to renew its CE marking.

DETAILED DESCRIPTION:
The LeMaitre Cardial Dialine® II Vascular Prostheses (Dialine II) is a knitted PET (Polyethylene Terephthalate) graft manufactured with multifilament yarns and impregnated with bovine origin collagen to achieve a strong and dilatation resistant graft, which eliminates the preclotting step. The bovine collagen is then gradually resorbed by the patient. The Dialine II comes with black guide lines and crimped construction to facilitate implantation.

Other design features include:

* Thin wall design (0.50+/-0.12mm) with excellent conformability
* Special impregnation process for maximum leakage resistance
* Water permeability < 10 ml/cm2/min

The Dialine II is indicated for replacement or bypass procedures in aneurysmal and/or occlusive diseases of the abdominal aorta or peripheral arteries. The Dialine II is also indicated for arterial reconstruction in patients requiring systemic heparinization. The unique collagen impregnation results in exceptional resistance to leakage, even under systemic heparinization.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ≥ 18 years of age
* Subject who has undergone surgical treatment for the replacement or bypass in aneurysmal and/or occlusive diseases and for arterial reconstruction in patients requiring systemic heparinization with LeMaitre Cardial Dialine II (between 01JAN2010 and 31JUL2016).

Exclusion Criteria:

* Co-morbidity that in the discretion of the investigator might confound the results.
* Patient operated on with a Dialine II Vascular prosthesis in conditions where it is connected with another one and that will make impossible to attribute the complication in the case it occurs
* Infection that may affect the safety or the efficacity of the prothesis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects who have undergone surgical treatment for the replacement or bypass in aneurysmal and/or occlusive diseases and for arterial reconstruction in patients requiring systemic heparinization with LeMaitre Cardial Dialine II.
Sampling Method: Non-Probability Sample
Enrollment: 262 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Primary patency of the prothesis | 1 year
Occurence of serious adverse events | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nabil CHAKFE, PUPH-MD-PhD, Principal Investigator — Hôpitaux Universitaires de Strasbourg - GEPROVAS
Locations (1):
- GEPROVAS, Strasbourg, Bas-Rhin, France

IPD SHARING:
Plan to Share IPD: Undecided